CLINICAL TRIAL: NCT02660944
Title: A Phase 2a, Double-blind, Placebo-Controlled Study of RSLV-132 in Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: A Phase 2a of RSLV-132 in Subjects With Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Resolve Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 132-03
Record Dates: First submitted 2016-01-16; First posted 2016-01-21 (Estimated); Results first posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — RSLV-132

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RSLV-132 (Experimental): 10 mg/kg RSLV-132
  Interventions: Drug: RSLV-132
- Placebo (Placebo Comparator): Saline placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RSLV-132 — RNase-Fc fusion protein
  Arms: RSLV-132
Drug: Placebo — Saline placebo
  Arms: Placebo

SUMMARY:
This study evaluates the impact of 13 bi-weekly intravenous infusions of RSLV-132 on the cutaneous manifestations in subjects with systemic lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

* CLASI score greater than or equal to 10 at Baseline
* Positive for one or more RNA autoantibodies

Exclusion Criteria:

1. severe, active central nervous system (CNS) involvement at Screening;
2. severe renal involvement at Screening (urine protein/creatinine ratio of >200 mg/mmol, or an estimated creatinine clearance of <30 mL/min);
3. use of cyclophosphamide within 3 months of the Baseline visit;
4. use of rituximab within 6 months of the Baseline visit;
5. use of belimumab within 3 months of the Baseline visit;
6. use of background medications within 1 month of Baseline in excess of: i. mycophenolate mofetil > 3 g/day; ii. azathioprine > 200 mg/day; iii. methotrexate > 25 mg/day; iv. hydroxychloroquine > 400 mg/day; v. prednisone (or equivalent) > 15 mg/day;
7. use of an intravenous steroid "pulse" within 2 months of Baseline;
8. use of an intramuscular steroid injection within 1 month of Baseline;
9. change in SLE medications within 1 month of Baseline;
10. the presence of a clinically significant infection in the judgement of the Investigator within seven days prior to the receipt of the first dose of study drug;
11. positive viral load test for hepatitis B, C, or HIV at Screening;
12. participation in another clinical trial with receipt of an investigational product within 3 months or 5 half- lives, of last administration (whichever is longer) from Baseline;
13. positive pregnancy test at Screening or at Baseline;
14. female subjects currently breast feeding at Baseline;
15. inability or unwillingness to comply with protocol-specified procedures which, in the opinion of the Investigator, would make the subject unsuitable for study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-01-03 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Posada, Ph.D., Study Chair — Resolve Therapeutics
Locations (16):
- United States (16):
  - TriWest Research Associates, El Cajon, California
  - University of California San Diego, La Jolla, California
  - Valerius Research Center, Los Alamitos, California
  - Wallace Rheumatic Study Center, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Clinical Research of West Florida, Clearwater, Florida
  - Center for Rheumatology, Immunology and Arthritis, Fort Lauderdale, Florida
  - Alper Research, Naples, Florida
  - Northwell Health/ Division of Rheumatology, Great Neck, New York
  - Feinstein Institute for Medical Research, Manhasset, New York
  - DJL Clinical Research, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Metroplex Clinical Research Center, Dallas, Texas
  - Accurate Clinical Research, Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RSLV-132 | Placebo
Started | 42 | 22
Completed | 25 | 12
Not Completed | 17 | 10
Not completed — Adverse Event | 3 | 4
Not completed — Physician Decision | 3 | 1
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Lost to Follow-up | 4 | 1
Not completed — Subject schedule | 0 | 1
Not completed — Exclusion criteria met | 2 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | RSLV-132 | Placebo | Total
Number analyzed (Participants) | 42 | 22 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (12.8) | 45.2 (11.6) | 45.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 22 | 61
  Male | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 4 | 17
  Not Hispanic or Latino | 29 | 18 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 11 | 27
  White | 22 | 11 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 32 | 22 | 54
CLASI Activity Total Score [Mean (Standard Deviation); unit: Score on a scale] — Mean Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Activity Score. The CLASI is a single-page tool that separately quantifies disease activity and damage. For the activity score, points are given for the presence of erythema, scale, mucous membrane lesions, recent hair loss, and inflammatory alopecia. The total score represents the sum of the individual scores and ranges from 0 to 70. Higher scores are awarded for more severe manifestations.
  Score on a scale | 24.1 (9.9) | 22.4 (7.9) | 23.5 (9.2)
Oral corticosteroid dose [Count of Participants; unit: Participants]
  0 | 20 | 7 | 27
  >0 and less than or equal to 7.5 mg/kg | 6 | 5 | 11
  >7.5 | 16 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: Mean Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Improvement Compared to Placebo.
Description: Mean change from baseline (from baseline to Day 85; or baseline to Day 169) in CLASI activity scores (Last Observation Carried Forward [LOCF] post censoring values).
  The CLASI is a single-page tool that separately quantifies disease activity and damage. For the activity score, points are given for the presence of erythema, scale, mucous membrane lesions, recent hair loss, and inflammatory alopecia. The total score represents the sum of the individual scores and ranges from 0 to 70. Higher scores are awarded for more severe manifestations.
Time Frame: Baseline and Days 29, 57, 85, 99, 113, 127, 141, 155, 169
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | RSLV-132 | Placebo
Number analyzed (Participants) | 42 | 22
Scores on a scale
  Day 85 | -6.2 (6.7) | -6.5 (6.2)
  Day 169 | -6.2 (8.5) | -5.7 (7.0)
Statistical Analysis 1: Comparison: RSLV-132 vs Placebo; Change from baseline at Day 85 RSLV-132 versus placebo; Test type: Superiority — Two-sample t-test with Satterthwaite approximation; p = 0.845, t-test, 2 sided; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-3.42 to 4.15]
Statistical Analysis 2: Comparison: RSLV-132 vs Placebo; Change from baseline at Day 169 RSLV-132 versus placebo; Test type: Superiority — Two-sample t-test with Satterthwaite approximation; p = 0.818, t-test, 2 sided; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-4.66 to 3.70]

2. Secondary Outcome: Percentage of Participants Achieving a 50% Improvement in CLASI Activity Score
Description: Percentage of participants achieving a 50% improvement in CLASI activity score at Day 85 and Day 169 (LOCF post censoring due to use of exclusionary medications)
Time Frame: Baseline and Days 29, 57, 85, 99, 113, 127, 141, 155, 169
Population: On Day 169, a post hoc exploratory subgroup analysis was performed on participants with severe CLASI and severe SLE Disease Activity Index (SLEDAI-2K) scores at baseline. The SLEDAI-2K is a clinical index for the assessment of lupus disease activity in the previous 30 days. It consists of 24 weighted clinical and laboratory variables of nine organ systems. Scores of the descriptors range from 1 to 8, the total possible score is 105. A higher score indicates more severe disease.
Measure: Count of Participants; unit: Participants
Arm/Group | RSLV-132 | Placebo
Number analyzed (Participants) | 42 | 22
Participants
  Day 85: number analyzed (Participants) | 37 | 17
  Day 85 | 11 | 2
  Day 169 All Participants | 14 | 5
  Day 169 Participants with Severe CLASI >/=21: number analyzed (Participants) | 18 | 12
  Day 169 Participants with Severe CLASI >/=21 | 7 | 3
  Day 169 Participants with Severe SLEDAI >/=9: number analyzed (Participants) | 13 | 9
  Day 169 Participants with Severe SLEDAI >/=9 | 4 | 1

3. Post Hoc Outcome: Percentage of Participants With SRI-4 Response
Description: Percentage of participants with an Systemic Lupus Erythematous Responder Index (SRI) 4 response on Day 169. This is a composite responder index incorporating the British Isles Lupus Assessment Group (BILAG) 2004, SLEDAI-2K and Physician Global Assessment (PGA) responses. The BILAG-2004 index, an organ-based transitional activity instrument, provides disease activity scorings across nine organ systems (constitutional, mucocutaneous, neuropsychiatry, musculoskeletal, cardiorespiratory, gastrointestinal, ophthalmic, renal and hematological) on an ordinal scale (A to E) based on the physician's intention-to-treat premise. Grade A represents the most active and Grade E the least active disease. The Physician's Global Assessment is measured on a 0 to 100 mm scale with score 0 to be No Disease Activity and score 100 to be the most Severe Disease Activity.
Time Frame: Baseline and Day 169
Population: A subgroup analysis was also performed on participants with severe CLASI and severe SLEDAI scores
Measure: Count of Participants; unit: Participants
Arm/Group | RSLV-132 | Placebo
Number analyzed (Participants) | 42 | 22
Participants
  Day 169 All participants: number analyzed (Participants) | 39 | 20
  Day 169 All participants | 11 | 7
  Day 169 Participants with Severe CLASI >/=21: number analyzed (Participants) | 18 | 12
  Day 169 Participants with Severe CLASI >/=21 | 7 | 1
  Day 169 Participants with Severe SLEDAI >/=9: number analyzed (Participants) | 13 | 9
  Day 169 Participants with Severe SLEDAI >/=9 | 8 | 4

4. Post Hoc Outcome: Percentage of Participants With a British Isles Lupus Assessment Group-based Composite Lupus Assessment (BICLA) Response
Description: Percentage of participants with a BICLA response on Day 169. This is a composite responder index incorporating the BILAG-2004, SLEDAI-2K and PGA responses. The BILAG-2004 index, an organ-based transitional activity instrument, provides disease activity scorings across nine organ systems (constitutional, mucocutaneous, neuropsychiatry, musculoskeletal, cardiorespiratory, gastrointestinal, ophthalmic, renal and hematological) on an ordinal scale (A to E) based on the physician's intention-to-treat premise. Grade A represents the most active and Grade E the least active disease. The PGA is measured on a 0 to 100 mm scale with score 0 to be No Disease Activity and score 100 to be the most Severe Disease Activity.
Time Frame: Baseline and Day 169
Population: A subgroup analysis was also performed on participants with severe CLASI and severe SLEDAI scores
Measure: Count of Participants; unit: Participants
Arm/Group | RSLV-132 | Placebo
Number analyzed (Participants) | 42 | 22
Participants
  Day 169 All Participants: number analyzed (Participants) | 39 | 20
  Day 169 All Participants | 10 | 4
  Day 169 Participants with Severe CLASI >/=21: number analyzed (Participants) | 18 | 12
  Day 169 Participants with Severe CLASI >/=21 | 5 | 1
  Day 169 Participants with Severe SLEDAI >/=9: number analyzed (Participants) | 13 | 9
  Day 169 Participants with Severe SLEDAI >/=9 | 4 | 1

ADVERSE EVENTS:
Time Frame: 215 days
Description: Treatment emergent adverse events are summarized
Arm/Group | RSLV-132 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/22
Serious Adverse Events (participants affected / at risk) | 3/42 | 5/22
Other Adverse Events (participants affected / at risk) | 36/42 | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSLV-132 (N=42) | Placebo (N=22)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Escherichia Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Flank Pain (Infections and infestations) | 0 (0) | 1 (1)
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Cutaneous Lupus Erythematosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSLV-132 (N=42) | Placebo (N=22)
Hypertension (Vascular disorders) | 6 (6) | 4 (4)
Headache (Nervous system disorders) | 6 (7) | 3 (4)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (3)
Urinary Tract Infection (Infections and infestations) | 4 (5) | 4 (4)
Cutaneous Lupus Erythematosus (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Sinusitis (Infections and infestations) | 4 (4) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (4) | 4 (5)
Proteinuria (Renal and urinary disorders) | 3 (4) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT02660944/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT02660944/SAP_001.pdf